CLINICAL TRIAL: NCT04581681
Title: Group Cognitive Behaviour Therapy for Perinatal Anxiety: a Randomized Controlled Trial
Brief Title: Group Cognitive Behavioural Therapy (CBT) for Perinatal Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Gillian Alcolado, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2020:095
Record Dates: First submitted 2020-09-22; First posted 2020-10-09 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-06

CONDITIONS: Perinatal Anxiety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group CBT for Perinatal Anxiety (Experimental): Using cognitive-behavioural therapy principles, this group therapy is intended to treat perinatal anxiety.
  Interventions: Behavioral: Group Cognitive Behaviour Therapy for Perinatal Anxiety (CBT-PA)
- Waitlist Control (Active Comparator): This is a control condition in which patients are randomly assigned to the waitlist control condition before receiving the treatment.
  Interventions: Other: No treatment (waitlist control)

INTERVENTIONS:
Behavioral: Group Cognitive Behaviour Therapy for Perinatal Anxiety (CBT-PA) — The 6-session group CBT intervention for perinatal anxiety has been formalized with session guides for the facilitators and a workbook, "Overcoming Anxiety in Pregnancy and Postpartum" (Furer & Reynolds, 2015), developed by members of our Anxiety Disorders Clinic. There are 6 core modules covered over the 6 treatment sessions, including: (1) Understanding anxiety during pregnancy and postpartum, (2) self-care, (3) setting goals and facing fears, (4) nurturing the developing relationship with baby, (5) coping with negative thoughts and worries, and (6) relapse prevention. Content is based on general principles of CBT for anxiety but specific themes and examples are geared towards the pregnancy and postpartum periods. Distorted cognitions are also explored, with an additional focus on beliefs about motherhood and perfectionism. Due to the COVID-19 pandemic, the intervention will be conducted via a hospital-approved video-conferencing platform.
  Arms: Group CBT for Perinatal Anxiety
Other: No treatment (waitlist control) — Patients in this condition are randomly assigned to a waitlist control condition before receiving treatment.
  Arms: Waitlist Control

SUMMARY:
Our previous pilot study (N = 40) suggested that group Cognitive Behaviour Therapy for perinatal anxiety (CBT-PA) significantly reduces symptoms of anxiety and depression from pre- to post- intervention. CBT-PA is based on the general principles of CBT but specific themes and examples are geared towards pregnancy and postpartum periods. The 6-week treatment protocol addresses: (1) understanding anxiety during pregnancy and postpartum, (2) self-care, (3) setting goals and facing fears, (4) nurturing the developing relationship with baby, (5) coping with negative thoughts and worries, and (6) relapse prevention. This intervention and all assessment interviews will be conducted via a hospital-approved video-conferencing platform. All assessment questionnaires will be completed on SurveyGizmo. The objectives of the present study are: (1) to replicate these findings of the pilot study in a larger sample (N = 58) in a randomized controlled trial (RCT), (2) compare the effectiveness of CBT-PA to a control treatment (waitlist control), (3) evaluate the durability of treatment gains at 1-month and 3-months after the conclusion of treatment, (4) evaluate patient preferences in terms of the relevance and the acceptability of the CBT-PA protocol, (5) examine whether the degree of childbirth stress impacts patient response to CBT-PA to inform future refinements to the treatment, and (6) determine whether CBT-PA improves maternal efficacy and attachment with baby. This research is being conducted because many women suffer from perinatal anxiety and have difficulty accessing services in a timely manner. It is the hope that the findings of this study will have clinical significance in terms of providing additional support for CBT as an effective treatment for perinatal anxiety. It is the hope that this treatment will have mental and physical health benefits for the mothers directly, as well as mental and physical health benefits to their fetuses and infants.

ELIGIBILITY:
Inclusion Criteria:

* Adult over the age of 18 years living in the province of Manitoba, Canada.
* Must be pregnant or within 12 months postpartum.
* Women must also meet criteria for at least one anxiety disorder or related disorder (i.e., generalized anxiety disorder, social anxiety disorder, panic disorder with or without agoraphobia, obsessive-compulsive disorder, or posttraumatic stress disorder).

Exclusion Criteria:

* Primary perinatal depression
* Active suicidality and/or homicidality
* Active psychosis, manic, or a substance use disorder that would interfere with participation in treatment.
* Women also must not be receiving concurrent psychotherapy
* If on medication, must not have made any medication changes in the 6 weeks prior to beginning participation in our study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Perceived Stress Scale | Pre-treatment (intake assessment); immediately post-treatment; 1- and 3-month follow-ups; and weekly during treatment up to 6 weeks
  This is a 10-item self-report measure that assesses the extent to which one's life is appraised as stressful. Scores can range from 0 to 40, with higher scores indicating higher levels of perceived stress.
Changes in scores on the Perinatal Anxiety Screening Scale | Pre-treatment (intake assessment); immediately post-treatment; 1- and 3-month follow-ups; and weekly during treatment, up to 6 weeks
  This is a 31-item self-report measure assessing symptoms of anxiety during the perinatal period. Scores on this measure can range from 0 to 93, with higher scores indicating higher levels of anxiety. It will be used in the current investigation to examine changes in anxiety symptoms across time.

SECONDARY OUTCOMES:
Change in scores on the The Edinburgh Postnatal Depression Scale | Pre-treatment (intake assessment), immediately post-treatment; 1-month follow-up; 3-month follow-up; and weekly during treatment, up to 6 weeks
  10-item self-report measure assessing symptoms of postnatal depression on a 0 to 3 scale. Scores can range from 0 to 30, with higher scores indicating higher levels of postnatal depression.
Change in scores on the Maternal Antenatal Attachment Scale | Pre-treatment (intake assessment), immediately post-treatment, 1-month follow-up, 3-month follow-up
  This is a 19-item self-report measure that assesses maternal attachment towards her unborn baby in the antenatal period. This measure will be administered to women who are participating in the study during the prenatal period. Scores range from 19 to 95, with higher scores indicating a higher level of attachment to the fetus.
Change in scores on the Maternal Efficacy Questionnaire | Pre-treatment (intake assessment), immediately post-treatment, 1-month follow-up, 3-month follow-up
  This is a 10-item self-report measure that assesses a mother's perception of her own parenting competence. Scores on this measure range from 10 to 40, with higher scores indicating higher levels of self-efficacy.
Change in scores on the Maternal Postnatal Attachment Scale | Pre-treatment (intake assessment), immediately post-treatment, 1-month follow-up, 3-month follow-up
  This is a 19-item self-report measure that assesses maternal attachment towards her infant during the postnatal period. This measure will be administered to women who are participating in the study during the postpartum period. Higher scores indicate higher levels of attachment to baby.
Post-Delivery Perceived Stress Inventory | Pre-treatment (intake assessment)
  This is a 29-item self-report measure of the degree of stress experienced as a result of the birth experience specifically. The PPSI will be administered at the intake assessment to postpartum women. Scores range from 0 to 116, with higher scores indicating higher levels of perceived stress.
The Treatment Acceptability/Adherence Scale | Pre-treatment (at the outset of treatment)
  This is a self-report measure of treatment acceptability. It will be administered at treatment outset to determine the perceived acceptability of the treatment to participants. Scores range from 7 to 70, with higher scores indicating higher levels of treatment acceptability.
The Treatment Satisfaction Measure | Immediately post-treatment
  This measure was developed for use in our clinic to evaluate patient impressions of treatment. Four items regarding the helpfulness of the sessions, the group aspect, the workbook, and the focus on perinatal issues are rated on a 5-point scale (i.e., from "very helpful" to "not at all helpful"). Two additional yes/no questions are included, regarding whether participants would recommend the program to other perinatal women and whether they themselves would participate in the group again if needed. Two final open-ended questions are included regarding what patients liked about group, and any suggestions they would have for changes to future groups.
Change in scores on the The Hamilton Anxiety Rating Scale | Pre-treatment; immediately post-treatment; 1-month post-treatment; 3-months post-treatment
  A 14-item clinician-administered interview scale used to assess the severity of anxiety symptoms. It will be used in the present study to examine changes in anxiety symptoms from pre- to post-treatment. Scores can range from 0 to 30, with higher scores indicating greater anxiety severity.
The Homework Checklist | From group treatment session two, up to five weeks.
  A list of all homework assignments from each session. Participants will complete the list at each session regarding the previous week's homework assignments, whether they worked on each element, for how long, and any comments they might have.
The Treatment Protocol Adherence Checklist | Completed by group leaders weekly, up to 6 weeks.
  A checklist copy of the group leader's guide to each session, with a spot to check off if each element was covered, and open-ended questions regarding deviations from the protocol; and other session occurrences of note.
The Coronavirus Stressor Survey | Pre-treatment (intake assessment)
  A 10-item survey that asks about the impact of the coronavirus pandemic on the lives of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No